CLINICAL TRIAL: NCT06023264
Title: Randomized, Open Clinical Trial to Evaluate the Effect of Dry Needling on the Temporomandibular Joint in Subjects Who Have Suffered a Whiplash as a Result of a Traffic Accident
Brief Title: Evaluate the Effect of Dry Needling on the Temporomandibular Joint in Subjects Who Have Suffered a Whiplash as a Result of a Traffic Accident
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03916375G
Record Dates: First submitted 2023-08-17; First posted 2023-09-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-08

CONDITIONS: Whiplash; Temporomandibular Joint Pain; Dry Needling Technique
MeSH Terms: conditions — Whiplash Injuries | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- dry needle (Experimental)
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — It is a minimally invasive treatment modality. Its effectiveness has been confirmed in numerous studies. It consists of applying an antiseptic in the puncture area and inserting the needle in the required aseptic conditions. During puncture, the patient's physical response is observed at all times, in order to control the local spasmodic responses in each muscle. After applying the technique, we assessed jaw pain, mouth opening, and the appearance of headaches. The adverse effects of the technique are the following: pain after puncture (1.7%), local bleeding at the puncture site (6.1%) and syncopal responses (0.7%).
  Arms: dry needle

SUMMARY:
The transportation industry is growing rapidly and the most popular mode is overland by road. Traffic accidents are the most direct and serious risk to the lives of Western people. A large number of traffic accidents occur on the roads each year, especially those caused by motor vehicles on motorways and urban ring roads, often resulting in massive loss of life. According to the World Health Organization (WHO), 1.35 million people die each year worldwide.

Whiplash is the most common injury in motor vehicle collisions, affecting 83% of injured people.

The temporomandibular joint (TMJ) is one of the most complex joints in the human body, since in addition to performing functions in dental occlusion, it does so in the neuromuscular system.

Due to the relationship of the neck with the mandible, the main objective of the study is to determine if there is an improvement in pain and functional limitation in general by applying the dry needling technique in the temporomandibular joint musculature.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered a traffic accident
* Having suffered a subsequent collision
* Having been diagnosed with whiplash in the hospital ''Fundación Jiménez Díaz (FJD)´´ emergency room in the first 72 hours after the collision.
* Age between 18-45 years, to avoid osteoarthritis and other degenerative problems.
* Minimum 3 in temporomandibular joint (TMJ) according to Visual Analog Scale (VAS)
* Consent to participate

Exclusion Criteria:

* Temporomandibular joint (TMJ) or craniofacial surgeries
* Spinal surgery
* Direct trauma in temporomandibular joint (TMJ) or prior to the accident
* Botox, silicones or any type of cosmetic surgery in the facial region.
* Problems of migraines and tension headaches (pre-accident)
* Any degenerative musculoskeletal disease (fibromyalgia, rheumatoid arthritis, osteoarthritis)
* Fear of needles
* Any neurological disorder (trigeminal neuralgia, epilepsy)
* Pregnancy
* Uncontrolled vascular or metabolic problems

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Age | Visit 1 (First day of treatment)
  Years (Demographic variables)
Gender | Visit 1 (First day of treatment)
  Male, Female, Does not answer (Demographic variables)
Weight | Visit 1 (First day of treatment)
  Kilograms (Demographic variables)
Height | Visit 1 (First day of treatment)
  Meters (Demographic variables)
Mouth opening | Visit 1(First day of treatment) and Visit 2 (One week after visit 1)
  Millimeters (Basal conditions)
Jaw pain | Visit 1(First day of treatment) and Visit 2 (One week after visit 1)
  Visual Analog Scale (VAS) 1-10 (Basal conditions)
Headache | Visit 1(First day of treatment) and Visit 2 (One week after visit 1)
  Visual Analog Scale (VAS) 1-10 (Basal conditions)
Joint clicking | Visit 1(First day of treatment) and Visit 2 (One week after visit 1)
  Yes/No (Basal conditions)
Pressure masseter, pterygoid, and temporalis | Visit 1 (First day of treatment)
  Determine pressure in kg in the masseter, temporal, and pterygoid muscles with an algometer to obtain 5/10 in Visual Analog Scale (VAS) to all participants
Pain masseter, pterygoid, and temporalis | Visit 1(First day of treatment) and Visit 2 (One week after visit 1)
  Obtain pain from 1 to 10 in the masseter, temporal, and pterygoid muscles according to the Visual Analog Scale (VAS) after applying the pressure obtained with the algometer in the previous step. *Patients in the experimental group are evaluated 10 minutes after the application of dry needling

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Universidad de Alcalá de Henares, Madrid
  - Patricia Recio Ramos, Madrid

IPD SHARING:
Plan to Share IPD: No